CLINICAL TRIAL: NCT07091396
Title: Enhancing Functional Recovery With Home-based Transcranial Direct Current Stimulation (tDCS) in Patients With Stroke, Neurodegeneration and Brain Tumors
Brief Title: Home Transcranial Direct Current Stimulation (tDCS) to Enhance Functional Recovery
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Zafer Keser, Principal Investigator, Mayo Clinic
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 24-006350
Record Dates: First submitted 2025-07-17; First posted 2025-07-29 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Stroke; Neurodegeneration; Brain Tumor
Keywords: Transcranial Direct Current Stimulation (TDCS)
MeSH Terms: conditions — Stroke; Nerve Degeneration; Brain Neoplasms

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (4):
- Home-Based Treatment: Active Stimulation, Then Sham Stimulation (Experimental): Subjects will first receive active tDCS, plus home activity based cognitive-linguistic therapy then they will cross over to the home-based sham treatment arm after a 4-8-week washout period.
  Interventions: Device: Soterix® tDCS - Home treatment; Behavioral: Cognitive-linguistic therapy
- Home-Based Treatment: Sham Stimulation, Then Active Stimulation (Experimental): Subjects will first receive sham tDCS, plus home activity based cognitive-linguistic therapy then they will cross over to the home-based active treatment arm after a 4-8-week washout period.
  Interventions: Device: Soterix® tDCS - Home treatment; Behavioral: Cognitive-linguistic therapy
- Lab-Based Treatment: Active Stimulation, Then Sham Stimulation (Experimental): Subjects will be seen in person to first receive active tDCS for 12 sessions over 4 weeks, and cross-over to the lab-based sham treatment arm after an 8 week washout period.
  Interventions: Device: Soterix® tDCS - Lab treatment
- Lab-Based Treatment: Sham Stimulation, Then Active Stimulation (Experimental): Subjects will be seen in person to first receive sham tDCS for 12 sessions over 4 weeks, and cross-over to the lab-based active treatment arm after an 8 week washout period.
  Interventions: Device: Soterix® tDCS - Lab treatment

INTERVENTIONS:
Device: Soterix® tDCS - Home treatment — Participants will receive transcranial direct current stimulation (tDCS) via the Soterix device at an intensity of 2 mA for 20 minutes per session, with slow ramp-up and ramp-down of the current.
  Each participant will be asked to perform tDCS on weekdays for two-weeks (10 sessions total) or every other weekday for four weeks (12 sessions). The research team will decide on a number of therapy sessions depending on the patient's baseline condition and tolerance. Patients who receive 10 sessions of therapy over two weeks will have 4 weeks of washout. Patients who receive 12 sessions over four weeks will have 8 weeks of washout.
  Arms: Home-Based Treatment: Active Stimulation, Then Sham Stimulation; Home-Based Treatment: Sham Stimulation, Then Active Stimulation
Behavioral: Cognitive-linguistic therapy — Participants will be instructed to perform home activity based cognitive-linguistic task-based exercises. Each participant will be asked to perform tDCS concurrently with individualized activity based cognitive-linguistic therapy on weekdays for two-weeks (10 sessions total) or every other weekday for four weeks (12 sessions)
  Arms: Home-Based Treatment: Active Stimulation, Then Sham Stimulation; Home-Based Treatment: Sham Stimulation, Then Active Stimulation
Device: Soterix® tDCS - Lab treatment — Participants will receive transcranial direct current stimulation (tDCS) in person, via the same Soterix device the home based participants will use at an intensity of 2 mA for 20 minutes per session, with slow ramp-up and ramp-down of the current. They will undergo 12 sessions over four weeks.
  Arms: Lab-Based Treatment: Active Stimulation, Then Sham Stimulation; Lab-Based Treatment: Sham Stimulation, Then Active Stimulation

SUMMARY:
The purpose of this study is to assess the feasibility of home-based Transcranial Direct Current Stimulation (tDCS) combined with a home activity based therapy program in patients with stroke, brain tumors or neurodegenerative conditions and to assess the efficacy of home-based tDCS combined with a home activity-based therapy program as an intervention to treat cognitive-linguistic impairments related to stroke, brain tumors, or neurodegenerative conditions and improve quality of life.

ELIGIBILITY:
Inclusion Criteria:

* At least 3 months after ischemic/hemorrhagic/anoxic stroke or 3 months after completion of cranial radiation or cranial surgery for treatment of primary or metastatic intracranial tumors or neurodegenerative conditions include, but are not limited to, primary progressive aphasia, corticobasal syndrome, progressive supranuclear palsy, Parkinson's disease, and Alzheimer's disease dementia.
* Expected survival >6 months
* Functional impairment in the domains of language and/or cognition affecting quality of life determined by PI.
* Have a legally authorized representative who is able to sign on their behalf in unable to consent for themselves (ex., individuals with aphasia).
* Have a legally authorized representative who is able to sign on their behalf in unable to consent for themselves (ex., individuals with aphasia).

Exclusion Criteria:

* Pregnancy
* Contraindication to tDCS, including metallic implanted objects.
* Medical instability or inability to cooperate during the study as assessed by the treating physician to participate in the study.
* Individuals with epilepsy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Estimated)
Dates: Start 2026-01-16 (Actual); Primary Completion 2030-12 (Estimated); Study Completion 2031-12 (Estimated)

PRIMARY OUTCOMES:
For patients with post-stroke cognitive impairment--Stricker Learning Span and Symbols Test | Baseline, 3 weeks, 12 weeks, 15 weeks, 24 weeks
  The Stricker Learning Span (SLS) is a computer-adaptive digital word list memory test specifically designed for remote assessment and self-administration on a web-based multi-device platform (Mayo Test Drive).
For patients with post-stroke language impairment--Mayo-developed web-based language | Baseline, 3 weeks, 12 weeks, 15 weeks, 24 weeks
  The exam includes a standard protocol including sentence and word repetition, standard reading passage, vowel prolongation, speech alternating motion rates , sequential motion rates, picture description, naming, and animal fluency

SECONDARY OUTCOMES:
For patients with post-stroke language impairment--Western Aphasia Battery-Revised Bedside Version | Baseline, 12 weeks, 24 weeks
  Western aphasia battery assesses linguistic skills most frequently affected by aphasia such as content, fluency, auditory Comprehension, repetition and naming, reading, writing.
Change in Visual Analogue Scale to Evaluate Fatigue Severity (VAS-F) | Baseline, 3 weeks, 12 weeks, 15 weeks, 24 weeks
  The Visual Analogue Scale to Evaluate Fatigue Severity (VAS-F) is an 18 item self-report scale measuring the subject's experience of fatigue. Each item asks respondents to place an "X," representing how they currently feel, along a visual analogue line that extends between two extremes. Total scores range from 0 - 198, lower scores indicating lower levels of fatigue and higher scores indicating greater levels of fatigue.
Change in Epworth Sleepiness Scale (ESS) | Baseline, 3 weeks, 12 weeks, 15 weeks, 24 weeks
  The Epworth sleepiness scale (ESS) is an 8-item questionnaire that measures daytime sleepiness in participants. Possible scores range from 0-24, with higher scores indicating a higher average sleep propensity in daily life, and a worse outcome.
Karolinska Sleepiness Scale (KSS) | 10 minutes before and after each treatment session
  The Karolinska Sleepiness Scale (KSS) is a 9-point scale quantifying an individual's perceived level of drowsiness, ranging from 1 (extremely alert) to 9 (very sleepy, great effort to keep awake, fighting sleep).
Communicative Participation Item Bank | Baseline, 12 weeks, 24 weeks
  For patients with aphasia, this test will be used to measure functional impairment for speech and language functions

CONTACTS AND LOCATIONS:
Overall Officials: Zafer Keser, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials